CLINICAL TRIAL: NCT05676541
Title: Effectiveness of an Adaptive, Complex Intervention to Enhance Care for Patients With Complex Multimorbidity in General Practice - a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Enhanced Care for Patients With Complex Multimorbidity in Primary Care
Acronym: MM600-DK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Research Unit of General Practice, Odense (Other); Research Unit for General Practice, Aarhus University (Other); Slagelse Hospital (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCopenhagen-MM600
Record Dates: First submitted 2022-12-16; First posted 2023-01-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Multimorbidity
MeSH Terms: interventions — Multimorbidity

STUDY DESIGN:
Intervention Model Description: Cluster randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Complex intervention to enhance care for patients with multimorbidity in general practice consisting of an extended overview consultation and supporting elements
- Control (No Intervention)

INTERVENTIONS:
Other: Complex intervention to enhance care for patients with multimorbidity in general practice consisting of an extended overview consultation and supporting elements — The intervention consists of 1) an extended overview consultation lasting 30-45 minutes in general practice, 2) access to cross-sectoral video conferences with secondary care specialists and 3) an instruction material for GPs on how to organize the intervention and 4) an adaptive toolbox to support elements in the intervention (not yet developed)
  Arms: Intervention

SUMMARY:
Introduction Patients living with a chronic disease often have more than one chronic condition, which is referred to as multimorbidity. Multimorbidity is associated with decreased quality of life, functional decline, polypharmacy, and increased healthcare utilization. Patients with multimorbidity often have a high symptom- and treatment burden, and have to attend multiple appointments, often at numerous locations, and comply with complex or even conflicting advice and drug regimens, resulting in an increased risk of depression and low quality of life. In Denmark, general practice is the key organizational setting in terms of offering people with complex multimorbidity integrated, longitudinal, patient-centered care. However, caring for patients with multimorbidity is a complex and time-consuming task and the organization of chronic care in general practice is organized around individual conditions.

Research question The objective of the study is to evaluate the effectiveness of a complex intervention consisting of a prolonged consultation and a strengthened cross-sectoral collaboration for patients with complex multimorbidity listed in participating practices on the patients' health-related quality of life, health and use of health-services.

Methods

Design:

A pragmatic, adaptive, cluster-randomized, non-blinded, parallel-group trial conducted in general practice in all regions in Denmark evaluating a complex intervention.

ELIGIBILITY:
Inclusion Criteria:

Adult (18 years or older) patients listed at participating GPs living in their own home with

* Two or more chronic conditions from two of ten diagnosis groups OR who were identified by the GP with complex multimorbidity (see box 1)
* At least one contact with secondary care in 2022 or 2023.
* Prescribed at least five prescription drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Needs-based quality of life measured with MMQ1 - PROM | 2 years
  The primary outcome is needs-based quality of life measured with MMQ1 (unpublished at present). The outcome consist of six unidimensional domains; physical capacity, worries, limitations in daily activities, social life, self-image and economy with a scale from 0-3 per item (sum scores differ due to differences in the number f items) We expect our intervention to be able to affect the three domains; worries, limitations in daily life and social life.
  We will consider a clinically significant improvement in at least one domain as a success.

SECONDARY OUTCOMES:
Treatment burden (MMQ1-TB) - PROM | 2 years
  Under validation. The PROM consists of six domains with response categories from 0-3.
  a high score means high burden (negative)
Patient-perceived patient-centeredness of consultations (PCC-GP) -PROM | 2 years
  Under validation, The PROM consists of eight domains with response categories from 0-3. a high score means high patient-centeredness (positive)
Mortality - registry-based | 2 years
  Number of deaths in each group per patient-years at risk
Hospitalizations - registry-based | 2 years
  Number of hospitalizations in each group in total and per patient-years at risk. Any admittance to the hospital counts regardless if it is planned or unplanned and regardless the duration.
Nursing home placement registry-based | 2 years
  Number of nursing home placements in each group in total and per patient year at risk
number of prescription medicines - registry-based | 2 years
  Number of prescription medicines per patient in each group (as a count regardless indication)
Polypharmacy - registry-based | 2 years
  Number of patients with polypharmacy (more than 5 prescription drugs) in each group
GP work satisfaction related to care for patients with multimorbidity - questionnaire | 2 years
  We have developed six items regarding work satisfaction/burden in relation to working with patients with MM in general practice. A clinically significant difference between the groups in at least one of the items will be considered a success.
GP burn-out - questionnaire | 2 years
  If we get access to the national GP burnout questionnaire data, we will use the data to report this outcome. But the outcome depends on the questionnaire being distributed at an appropriate time which is not currently yet planned.
Use of health services in general practice registry-based | 2 years
  This outcome combines all use of health services in general practice regardless contact form. It will be measured as number of contacts
Use of other primary care health services (such as private specialists and out-of-hours care) registry-based. | 2 years
  All contacts in primary care will be combined and the number of contacts compared between groups
Use of outpatient and other planned health services in secondary care (including new referrals), registry-based | 2 years
  All contacts in secondary care will be combined and the number of contacts compared between groups
Health service use in the municipalities - registry-based | 2 years
  All contacts in the municipalities regarding health and rehabilitation will be combined and the number of contacts compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- General practices in all of Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen HH, Willadsen TG, Prior A, Lyhnebeck AB, Waldorff FB, Holm A. Methods and baseline results of the Cohort of Health-Related Outcomes in Chronic Illness Care in General Practice in Denmark (CHRONIC-GP). BMJ Open. 2025 Nov 26;15(11):e103807. doi: 10.1136/bmjopen-2025-103807. PMID 41298265
- [Derived] Lyhnebeck AB, Holm A, Buhl SF, Bissenbakker KH, Kristensen JK, Moller A, Prior A, Kamper-Jorgensen Z, Bocher S, Kristensen M, Waagepetersen A, Dalsgaard AH, Siersma V, Brodersen JB; MM600 trial group. Measuring treatment burden related to general practice in patients with multimorbidity: development and validation of a PROM. Fam Med Community Health. 2025 Aug 17;13(3):e003378. doi: 10.1136/fmch-2025-003378. PMID 40819910
- [Derived] Holm A, Lyhnebeck AB, Buhl SF, Bissenbakker K, Kristensen JK, Moller A, Prior A, Kamper-Jorgensen Z, Bocher S, Kristensen MAT, Waagepetersen A, Dalsgaard AH, Siersma V, Guassora AD, Brodersen JB; on behalf MM600 trial group. Development of a PROM to measure patient-centredness in chronic care consultations in primary care. Health Qual Life Outcomes. 2025 Jan 8;23(1):4. doi: 10.1186/s12955-024-02327-x. PMID 39780227
- [Derived] Holm A, Lyhnebeck AB, Rozing M, Buhl SF, Willadsen TG, Prior A, Christiansen AL, Kristensen J, Andersen JS, Waldorff FB, Siersma V, Brodersen JB, Reventlow S; MM600 project team. Effectiveness of an adaptive, multifaceted intervention to enhance care for patients with complex multimorbidity in general practice: protocol for a pragmatic cluster randomised controlled trial (the MM600 trial). BMJ Open. 2024 Feb 2;14(2):e077441. doi: 10.1136/bmjopen-2023-077441. PMID 38309759